CLINICAL TRIAL: NCT01215877
Title: A Phase II Study of Tesetaxel in Subjects Previously Treated With Chemotherapy for Metastatic Transitional Cell Carcinoma of the Urothelium
Brief Title: Tesetaxel for Previously Treated Patients With Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOBL204
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2011-11

CONDITIONS: Carcinoma, Transitional Cell
Keywords: Bladder cancer; Previously treated patients; Tesetaxel; Oral taxane
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — tesetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel capsules orally once every 21 days; duration of therapy not to exceed 12 months
  In Cycle 1, a dose of 27 mg/m2 will be administered. In subsequent cycles,
  * the dose will be increased to 35 mg/m2 in Cycle 2 for subjects who did not have an ANC < 1,500/mm3, a platelet count < 100,000/mm3, or a Grade 3 (or higher grade) nonhematologic adverse event considered by the Investigator to be related to protocol therapy (excluding alopecia, nausea, and vomiting) in Cycle 1. The dose is not to exceed the dose of 35 mg/m2 in any cycle subsequent to Cycle 2.
  * for all other subjects, the dose administered in Cycle 1 (27 mg/m2) will be administered in all subsequent cycles.
  Other Names: DJ-927

SUMMARY:
The intravenously administered taxanes, docetaxel and paclitaxel, alone and in combination with other chemotherapy agents are active in patients with advanced and metastatic bladder cancer, and agents of this class are a promising treatment option for some patients.

Tesetaxel is an orally administered taxane that is in development as treatment for subjects with advanced cancers. This study is being conducted to determine the efficacy and safety of tesetaxel administered to patients previously treated with chemotherapy for progressive metastatic transitional cell carcinoma of the urothelium.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histologically confirmed diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis
* Measurable disease (revised RECIST; Version 1.1)
* Karnofsky performance status ≥ 60%
* Previously treated with not more than 1 doublet or triplet regimen and that regimen contained gemcitabine and a platinum agent
* Adequate bone marrow, hepatic, and renal function, as specified in the protocol
* At least 4 weeks and recovery from effects of prior surgery, prior radiotherapy, or other therapy with an approved or investigational agent
* Ability to swallow an oral solid-dosage form of medication

Exclusion Criteria:

* Known metastasis or symptoms of metastasis to the central nervous system
* Significant medical disease other than cancer
* Presence of neuropathy > Grade 1 (NCI CTC, Version 4.0)
* Prior treatment with a taxane or other tubulin-targeted agent (eg, indibulin) other than a vinca alkaloid
* Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Response rate (revised RECIST) | 12 months from date of first dose of study medication for last patient enrolled
  Proportion of patients with a confirmed complete or partial response

SECONDARY OUTCOMES:
≥ 3-month response rate | 12 months from date of first dose of study medication for last patient enrolled
  Proportion of patients with a confirmed complete or partial response ≥ 3 months in duration
Disease control rate | 12 months from date of first dose of study medication for last patient enrolled
  Proportion of patients with a confirmed complete or partial response of any duration or stable disease ≥ 3 months in duration
Durable response rate | 12 months from date of first dose of study medication for last patient enrolled
  Proportion of subjects with a confirmed complete or partial response ≥ 6 months in duration
Duration of response | 12 months from date of first dose of study medication for last patient enrolled
  Date when response criteria are first met to the date when progression is first documented
Time to progression | 12 months from date of first dose of study medication for last patient enrolled
  Date of first dose of study medication to the date when progression is first documented
Safety | Up to 30 days after the last dose of study medication for a specific patient
  Adverse events and clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Dean F Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- San Camillo Forlanini Hospital, Rome, Italy